CLINICAL TRIAL: NCT05307887
Title: Does Virtual Reality Technology Reduce Pain and Anxiety During Outpatient Hysteroscopy? A Randomised Controlled Trial
Brief Title: Does Virtual Reality Technology Reduce Pain and Anxiety During Outpatient Hysteroscopy?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Imperial College Healthcare NHS Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 21SM7296
Record Dates: First submitted 2022-03-24; First posted 2022-04-01 (Actual); Results first posted 2024-08-09 (Actual); Last update posted 2024-08-09 (Actual); Status verified 2024-03

CONDITIONS: Anxiety; Pain
MeSH Terms: conditions — Anxiety Disorders; Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Virtual Reality Technology (Experimental): Group receiving virtual reality technology in addition to standard therapy
  Interventions: Device: Sync VR Medical PICO G2 4K Virtual Reality Technology
- Standard Therapy Control Group (No Intervention)

INTERVENTIONS:
Device: Sync VR Medical PICO G2 4K Virtual Reality Technology — Virtual reality headset and software
  Arms: Virtual Reality Technology

SUMMARY:
Hysteroscopy is a common procedure where a camera attached to a thin scope is passed into the uterus via the vagina and cervix in order to obtain views of the inside of the uterus. Hysteroscopy is used for the diagnosis and management of a variety of benign and conditions as well as the diagnosis of uterine cancer. It can be performed under general anaesthetic or in an outpatient setting without formal anaesthetic. The latter has several advantages when compared to hysteroscopy with general anaesthesia as it avoids the additional risk of general anaesthesia, has a quicker recovery time, shorter hospital stay and reduced cost. However, women may experience discomfort or pain during an outpatient procedure and pain is one of the most common reasons for failure to complete the procedure.

The most appropriate way to manage pain and anxiety during outpatient hysteroscopy is not yet fully understood and conventional therapy, as recommended by the Royal College of Obstetricians and Gynaecologists, involves the use of simple pain killers taken prior to the procedure and sometimes local anaesthetic during the procedure. In recent years virtual reality software has been developed and used in a variety of different settings to alleviate pain and anxiety during medical procedures.

This study aims to investigate whether the use of virtual reality as an adjunct to conventional pain management can reduce anxiety and pain during outpatient hysteroscopy. The study will take the form of a randomised controlled trial at St Mary's hospital London. A randomly selected group of patients undergoing outpatient hysteroscopy with conventional management plus the addition of virtual reality software will be compared to a control group of patients undergoing the procedure with conventional management only.

DETAILED DESCRIPTION:
BACKGROUND Hysteroscopy is a common gynaecological procedure where a camera attached to a thin scope is passed into the uterus via the vagina and cervix in order to obtain views of the inside of the uterus. Hysteroscopy is used for the diagnosis and management of a variety of benign and conditions as well as the diagnosis of uterine cancer. It can be performed under general anaesthetic or in an outpatient setting without formal anaesthetic. The latter has several advantages when compared to hysteroscopy with general anaesthesia as it avoids the additional risk of general anaesthesia, has a quicker recovery time, shorter hospital stay and reduced cost. Outpatient hysteroscopy (OPH) is generally well tolerated although some women will experience significant pain and pain is one of the most common reasons for failure to complete the procedure. As pain is one of the leading reasons for procedure failure, finding ways to reduce pain and anxiety is of critical importance. The optimal method of controlling pain and anxiety during outpatient hysteroscopy is poorly understood and hotly debated. Conventional therapy, as recommended by the Royal College of Obstetricians and Gynaecologists, involves the use of simple pain killers taken prior to the procedure and sometimes local anaesthetic during the procedure if dilatation of the cervix is required (RCOG 2011).Virtual reality (VR) technology is a relatively new and promising technology which if used as a distraction technique, may be able to reduce pain and anxiety experienced from a wide range of medical procedures. Virtual reality (VR) is a human-computer interface that provides users with various physical sensations (e.g., visual, haptic, auditory) to increase realism in the virtual world (Seth et al. 2011). To date VR has been used in a wide variety of inpatient and outpatient clinical scenarios to reduce pain and anxiety including simple blood tests, ENT procedures and minor gynaecological procedures such as hysterosalpingograms (Chan et al 2018, Wang et al 2020 and Ahmadpoura et al 2019). However, currently, to the best of our knowledge, there is only one relatively small-scale trial investigating the use of VR in an outpatient hysteroscopy setting (Deo et al 2020) meaning further studies are urgently needed to clarify the situation.

RATIONALE FOR CURRENT STUDY The purpose of this study would be to determine if the use of VR technology can reduce pain and anxiety experienced by patients during outpatient hysteroscopy procedures when compared to standard pain management.

The optimal method of controlling pain and anxiety during outpatient hysteroscopy is poorly understood and there is a wide variation in clinical practice. This study aims to test whether VR technology could reduce pain and anxiety as a relatively simple and safe adjunct to conventional pain management. Although VR has been used in a variety of clinical settings to date, there is only one previous study investigating the use of VR in an outpatient hysteroscopy setting (Deo et al 2020). The rationale of this study would be to build upon this evidence by performing the first large scale adequately powered randomised control trial of the use of VR technology in this setting.The study team hypothesises that the use of VR technology will significantly improve pain and anxiety when compared to conventional pain management. Finding additional low risk ways of improving pain and anxiety during OPH is of critical importance in order to improve patient experience and the success rate of the procedure as pain is a major reason for unsuccessful OPH procedures.

2. STUDY OBJECTIVES

The primary objectives of this study are to determine if:

1. VR technology can reduce pain during outpatient hysteroscopy?
2. VR technology can reduce anxiety during outpatient hysteroscopy?

The secondary objectives of this study are to determine if:

1. The use of VR technology feasible during outpatient hysteroscopy?
2. The use of VR during outpatient hysteroscopy reduces the procedure failure rate?
3. The use of VR increases the outpatient hysteroscopy appointment time? STUDY DESIGN The study design is an unblinded randomised controlled trial. This study design was chosen as it will provide the best quality of evidence with reduced bias compared to other study designs. A randomised controlled trial is also very feasible in this scenario. Neither the researchers nor the participants will be blinded as to which study arm they are in, as it would be impractical to do so with a VR headset used in the intervention group. The study will be adequately powered with a power calculation based upon findings from previous studies, meaning at least 40 patients will be included in each arm (at least 80 patients in total).

Patients will be randomly allocated by computer allocation to either the intervention or the control group. The intervention group will undergo OPH with standard care plus the use of VR technology administered through a headset with the option of wearing headphones (at the patient's discretion) or having the accompanying sound played aloud. The control group will undergo outpatient hysteroscopy with standard care. Standard care in this unit is in line with the RGCOG guidelines and involves advising patients to take ibuprofen and/or paracetamol one hour prior to their procedure unless there are contraindications. Local anaesthetic intracervical block is used at the discretion of the operator and is usually used if dilatation of the cervix is required.

The primary outcome measure will be the reported NRS (numeric rating score) score which is validated score to assess pain and anxiety levels with values from 0-11. The patient will be asked to fill out the NRS score prior to the hysteroscopy and following the hysteroscopy prior to leaving the clinic.Secondary outcome measures will be length of procedure, complication rate, reported side effects, procedure completion, hysteroscopy findings and type of procedure performed (for example if purely diagnostic or if any operative procedures are performed).

Participants will be recruited from the general gynaecology clinics. Only patients who have already opted to undergo outpatient hysteroscopy will be invited to take part in the study and they will be made aware of the study at the time of the clinic appointment or shortly after. Interested parties will then be contacted by the research team to discuss the study in more detail at a time which is convenient for the patient. Written consent to enter the study will be sought from the participant in advance of their procedure and only after a full explanation has been given. The patient will be offered a study information leaflet. Whilst waiting for their hysteroscopy procedure, the patient will be offered a face-to-face appointment with a member of the research team to discuss the study and sign the written consent form if they wish to participate in the study. If it is more convenient for the patient, and to avoid unnecessary additional appointments for the patient, they may prefer to discuss the study and go through the consent by phone before confirming consent on the day of the procedure. Patients will have time to consider whether to take part in the study prior to their procedure day and will be informed that they can withdraw consent for participation in the study at any time. Participating or not participating in the study will have no effect on the timing of the outpatient hysteroscopy or the type of procedure performed. Patients will have the opportunity to choose which virtual reality scenario they wish to experience during the procedure (choice of 4 scenarios from beach, space, underwater and zen four seasons).

At the time of their hysteroscopy. The patient will fill out the pre-procedure NRS score prior to entering the hysteroscopy room. The patient will then enter the outpatient hysteroscopy room where there will be the hysteroscopy team consisting of the lead hysteroscopist and the assistant, and also a single member of the research team who will have taken the study consent from the patient prior to their procedure. Following discussion with the hysteroscopist as usual, the patient will prepare for the procedure and position themselves on the procedure couch. Once comfortable, the member of the research team will help the patient to put on the VR headset (See appendix 1), and if the patient wishes, headphones. The virtual reality software will then start running and is controlled by the research team member, the software will run for the length of the procedure. The hysteroscopy team will be preparing the equipment as the virtual reality software is running. The member of the research team will remain in the room throughout the procedure to troubleshoot any issues with the headset or software and if necessary to stop the VR program. Following completion of the procedure the patient will fill out a NRS score prior to going home.

The VR software involves breathing exercises, relaxing music and a distracting immersive walk through a virtual environment. The scenario will be started and subsequently controlled by a member of the research team operating a tablet device. The hysteroscopy team will perform the procedure in exactly the same way as they would normally and any clinical decisions regarding potential procedures such as polypectomy, discontinuing or proceeding with the hysteroscopy will be made by the hysteroscopy team along with the patient in the usual way without any input from the research team member.

Maintaining appropriate clinical hygiene is of critical importance as the same headset will be used for different patients. The headset can be easily and effectively cleaned between use and the manufacturer (VR medical) provides a recommended cleaning regimen which we will use for the trial. After use, the VR device and controller should be cleaned with a damp microfibre cloth and disinfectant wipe, both the parts that have been in contact with the skin and the headbands.

The timetable for the project is expected to run as follows. Three months for preparation and obtaining ethical approval. Recruitment is expected to start following this and we would expect to obtain the required number of participants by 3 months based on the average referral rate for outpatient hysteroscopy in the unit being 150 patients per month and a 20% study participation rate. Data analysis and preparing the final report would take a further 3 months.Results will be recorded onto a pseudoanonymised database. Information will be collected from patients notes and imaging reports. Each patient will be allocated a study number and for each the following will be recorded:Age Parity Symptoms and duration Past medical history and co-morbidities BMI Previous surgery Current medication and medication used within the last 6 months Pain NRS (numeric rating score) Anxiety NRS Length of hysteroscopy procedure Time in Outpatient Procedure room Procedure successfully completed (or not) and reason for failure if appropriate Complications Hysteroscopy findings Type of hysteroscopic procedure performed STUDY OUTCOME MEASURES The primary outcome measure will be the reported NRS (numeric rating score) score which is validated score to assess pain and anxiety levels with values from 0-11. The patient will be asked to fill out the NRS score prior to the hysteroscopy and following the hysteroscopy prior to leaving the clinic.Secondary outcome measures will be length of procedure, complication rate, reported side effects, procedure completion, hysteroscopy findings and type of procedure performed (for example if purely diagnostic or if any operative procedures are performed).

ELIGIBILITY:
Inclusion Criteria:

* 1. Age 18-70 2. Patients undergoing outpatient hysteroscopy for any indication 3. Capacity to give informed consent 4. Cognitive and linguistic ability sufficient to understand and fill out the NRS questionnaire.

Exclusion Criteria:

* 1. Epilepsy 2. Severe vertigo 3. Hearing impairment 4. Current facial injury /burn 5. Patients who have not given informed consent 6. Patients aged less than 18 or more than 70.

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 83 (Actual)
Dates: Start 2022-04-25 (Actual); Primary Completion 2022-10-11 (Actual); Study Completion 2022-10-11 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- St Mary's Hospital, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment was performed between April and October 2022 at St Mary's Hospital London gynaecology clinics.
Groups:
- Standard Therapy Control Group: Group receiving standard care including simple analgesia prior to procedure.
Period: Overall Study
Arm/Group | Virtual Reality Technology | Standard Therapy Control Group
Started | 41 | 42
Completed | 41 | 42
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Standard Therapy Control Group: Group receiving standard care
- Total: Total of all reporting groups
Arm/Group | Virtual Reality Technology | Standard Therapy Control Group | Total
Number analyzed (Participants) | 41 | 42 | 83
Age, Continuous [Mean (Standard Deviation); unit: years] | 47.8 (11.3) | 49.6 (11.3) | 48.7 (10.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 41 | 42 | 83
  Male | 0 | 0 | 0
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Parity [Mean (Standard Deviation); unit: pregnancies] | 0.9 (1.2) | 1.1 (1.4) | 1.1 (1.4)
Number of Post-menopausal Participants [Count of Participants; unit: Participants] — Number of post menopausal patients in each group with the menopause defined as absence of a menstrual period for 12 months or more.
  Participants | 16 | 17 | 33
Body mass index [Mean (Standard Deviation); unit: kg/m2] | 26.4 (6.2) | 26.8 (6.1) | 26.6 (6.1)
History of chronic pain [Count of Participants; unit: Participants] | 3 | 5 | 8
History of anxiety [Count of Participants; unit: Participants] | 2 | 5 | 7
Baseline anxiety levels [Mean (Standard Deviation); unit: units on a scale] — NRS score 0-10, with 0 being no anxiety and 10 being maximal anxiety.
  units on a scale | 4.0 (3.2) | 4.4 (3.0) | 4.2 (3.0)
Baseline pain level [Mean (Standard Deviation); unit: units on a scale] — NRS score 0-10, with 0 being no pain and 10 being maximal pain.
  units on a scale | 2.5 (2.9) | 2.5 (2.7) | 2.5 (2.8)
Preprocedure analgesia [Count of Participants; unit: Participants] | 33 | 37 | 70

OUTCOME MEASURES:

1. Primary Outcome: Reported Numeric Rating Score (NRS) Pain Score
Description: Self reported procedure related pain score (0-11 with higher numbers indicating increased pain).
Time Frame: Following completion of the procedure( within 20 minutes of completion).
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Virtual Reality Technology | Standard Therapy Control Group
Number analyzed (Participants) | 41 | 42
units on a scale | 3.73 (2.39) | 4.24 (3.07)

2. Primary Outcome: Reported Numeric Rating Score (NRS) Anxiety Score
Description: Self reported procedure related anxiety score (0-11 with higher numbers indicating higher anxiety levels).
Time Frame: Following completion of the procedure( within 20 minutes of completion).
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Virtual Reality Technology | Standard Therapy Control Group
Number analyzed (Participants) | 41 | 42
units on a scale | 3.29 (2.93) | 4.79 (3.38)

3. Secondary Outcome: Procedure Time
Description: Time taken to complete hysteroscopy procedure
Time Frame: From start to end of procedure
Measure: Mean (Standard Deviation); unit: minute
Arm/Group | Virtual Reality Technology | Standard Therapy Control Group
Number analyzed (Participants) | 41 | 42
minute | 9.5 (5) | 7.6 (3.7)

4. Secondary Outcome: Patient Pain Control Satisfaction
Description: Self reported procedure related satisfaction score (0-11 with higher numbers indicating higher patient satisfaction with the procedure).
Time Frame: Following completion of the procedure( within 20 minutes of completion).
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Virtual Reality Technology | Standard Therapy Control Group
Number analyzed (Participants) | 41 | 42
units on a scale | 8.4 (2.3) | 8.5 (2.4)

5. Secondary Outcome: Side Effects
Description: Any side effects or complications that occurred in each group.
Time Frame: during procedure
Measure: Count of Participants; unit: Participants
Arm/Group | Virtual Reality Technology | Standard Therapy Control Group
Number analyzed (Participants) | 41 | 42
Participants | 2 | 3

ADVERSE EVENTS:
Time Frame: Data was collected for each participant for the duration of their hysteroscopy procedure until they left the clinic (approx 30-60mins).
Arm/Group | Virtual Reality Technology | Standard Therapy Control Group
All-Cause Mortality (participants affected / at risk) | 0/41 | 0/42
Serious Adverse Events (participants affected / at risk) | 0/41 | 0/42
Other Adverse Events (participants affected / at risk) | 2/41 | 3/42
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Virtual Reality Technology (N=41) | Standard Therapy Control Group (N=42)
Nausea (Gastrointestinal disorders) | 2 (2) | 2 (2) — Felt nauseous during procedure.
vasovagal (Cardiac disorders) | 0 (0) | 1 (1) — Felt as if about to pass out, but no loss of consciousness experienced.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-02-14): https://cdn.clinicaltrials.gov/large-docs/87/NCT05307887/Prot_SAP_000.pdf